CLINICAL TRIAL: NCT06942065
Title: Clinical-randomized Study of the Influence of Rehabilitation Therapy Using Strength and Blood Flow Restriction Training on Muscular Fitness and Regeneration After Elective Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Alexander Franz, Dr. med., B.Sc., University Hospital, Bonn
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023_E
Record Dates: First submitted 2025-04-16; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Osteoarthritis (OA) of the Knee; Muscle Atrophy
MeSH Terms: conditions — Osteoarthritis; Muscular Atrophy | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Sham Comparator): Control sham condition which performed the exercise with a fixed pressure of 20mmHg
  Interventions: Procedure: Sham-BFR
- Blood Flow Restriction Group (Experimental): This intervention groups performed training on the operated limb with a BFR pressure corresponding to 60% of the individual limb occlusion pressure
  Interventions: Procedure: Blood Flow Restriction Training

INTERVENTIONS:
Procedure: Sham-BFR — The exercise protocol for the operated leg (with sham pressure of 20mmHg) consisted of four sets with 75 repetitions (reps) in total (1. Set: 30 reps, 2.-4. Set: 15 reps) with 30% of the individual one-repetition maximum for each exercise and were performed five times per week during the three-week outpatient rehabilitation.
  Arms: Control Group
Procedure: Blood Flow Restriction Training — The exercise protocol for the operated leg (with a BFR pressure of 60% of the LOP) consisted of four sets with 75 repetitions (reps) in total (1. Set: 30 reps, 2.-4. Set: 15 reps) with 30% of the individual one-repetition maximum for each exercise and were performed five times per week during the three-week outpatient rehabilitation.
  Arms: Blood Flow Restriction Group

SUMMARY:
The present study investigates the effects of blood flow restriction training on muscular recovery during out-patient rehabilitation after elective total knee arthroplasty

DETAILED DESCRIPTION:
The present study evaluated the impact of blood flow restriction training in the context of three-week outpatient rehabilitation following TKA, in accordance with the guidelines of the German Pension Insurance System. The in-rehabilitation and post-rehabilitation muscle status, strength, knee functionality, impairments in daily life and subjective pain perception were measured.

ELIGIBILITY:
Inclusion Criteria:

* Physical Fitness for Rehabilitation
* Primary TKA surgery
* BMI < 35

Exclusion Criteria:

* Sickle Cell Anemia
* Vascular Intervention on the lower extremities
* Open Wounds

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain | Pre- to 6 weeks Post Rehabilitation
  Postoperative Pain was assessed by visual analoge scale (0-100mm)
Muscle Strength | Pre- to 6 weeks Post Rehabilitation
  Isometric muscle strength was measured on a DDRobotec (Dynamic Devices AG, Zurich, Switzerland), a pneumatic, computer-controlled leg press

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Bonn, Bonn, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No